CLINICAL TRIAL: NCT05170295
Title: Noninvasive Monitoring of Cerebral Blood Flow Autoregulation
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.149
Record Dates: First submitted 2021-10-25; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Intracranial Pressure Increase; Cerebral Edema
Keywords: neuromonitoring; intracranial pressure (ICP); cerebral blood flow autoregulation; Rheoencephalography (REG); noninvasive neuromonitoring; cerebral edema; autoregulation; Cerebral Perfusion Pressure; Pressure reactivity index
MeSH Terms: conditions — Intracranial Hypertension; Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rheoencephalography (REG) shows promise as a method for noninvasive neuromonitoring, because it reflects cerebrovascular reactivity. This protocol will study clinical and technical conditions required to use REG. Additionally, our goal is to study noninvasive peripheral bioimpedance pulse waveforms in order to substitute invasive SAP. A previous study demonstrated that REG can be used to detect spreading depolarization (SD), the early sign of brain metabolic disturbance. SD can be measured invasively with DC EEG amplifiers only. Our goal is to create an automatic notification function for REG monitoring indicating change of clinical conditions.

DETAILED DESCRIPTION:
Neuromonitoring of patients with severe neurological illness are detailed elsewhere. In the setting of cerebral edema, ICP monitoring is a staple of neurocritical care. Pressure AR is an important hemodynamic mechanism that protects the brain against inappropriate fluctuations in CBF in the face of changing CPP. Both static and dynamic AR have been monitored in neurocritical care to aid prognostication and contribute to individualizing optimal CPP targets in patients. Theoretically, failure of cerebral AR is associated with poor outcomes in various acute neurological diseases. Continuous bedside monitoring of autoregulation is now feasible and should be considered as a part of multimodality monitoring including measurement of pressure reactivity. A previous study documented that REG (REGx) and ICP (PRx) has high correlation in order to detect the lower limit of CBF AR. The fundamental relationships between SAP, vessel tone, cerebral blood volume and ICP form the basis for the pressure reactivity index (PRx). PRx is analogous to other time domain AR indices and is calculated as the continuous correlation between thirty consecutive time-averaged (10 s) SAP and ICP values. A positive index (positive correlation) implies impaired passive CBF AR, while a negative index (inverse correlation) implies intact, active AR. The utility and feasibility of REG as a monitoring modality is previously demonstrated and validated as a reflection of cerebrovascular reactivity. The bioimpedance amplifier was used previously at Walter Reed Army Institute of Research (WRAIR) and Naval Medical Research Center (Silver Spring, MD); and has an FDA safety clearance. It is expected that REG can predict evolving vasospasm and expanding intracranial bleeding amongst several other clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Intact fronto-temporal area
* Intact lower arm area
* Clinical suspicion of elevated intracranial pressure

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve patients of Neurocritical Care Department with clinical suspicion of elevated intracranial pressure.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow Autoregulation (CBF AR) | through hospital admission, an average of 10 days
  Cerebral Blood Flow Autoregulation (CBF AR) will be analyzed based on noninvasive recordings (bioimpedance) by using a dedicated software for this purpose (part of ICM+ program, incorporated into a WRAIR-made software (DataLyser)). In this case CBF AR is called REGx.

SECONDARY OUTCOMES:
ICP Elevation | through hospital admission, an average of 10 days
  Morphological analysis of REG pulse waveform in order to detect ICP elevation, and establish the correlation between REGx and REG pulse waveform morphology.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cannizzaro, MD, Principal Investigator — Ochsner
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steiner LA, Andrews PJ. Monitoring the injured brain: ICP and CBF. Br J Anaesth. 2006 Jul;97(1):26-38. doi: 10.1093/bja/ael110. Epub 2006 May 12. PMID 16698860
- [Background] Donnelly J, Aries MJ, Czosnyka M. Further understanding of cerebral autoregulation at the bedside: possible implications for future therapy. Expert Rev Neurother. 2015 Feb;15(2):169-85. doi: 10.1586/14737175.2015.996552. PMID 25614952
- [Background] MCHENRY LC Jr. RHEOENCEPHALOGRAPHY: A CLINICAL APPRAISAL. Neurology. 1965 Jun;15:507-17. doi: 10.1212/wnl.15.6.507. No abstract available. PMID 14312772
- [Background] Traczewski W, Moskala M, Kruk D, Goscinski I, Szwabowska D, Polak J, Wielgosz K. The role of computerized rheoencephalography in the assessment of normal pressure hydrocephalus. J Neurotrauma. 2005 Jul;22(7):836-43. doi: 10.1089/neu.2005.22.836. PMID 16004585
- [Background] Bodo M, Simovic M, Pearce F, Ahmed A, Armonda R. Correlation of rheoencephalogram and intracranial pressure: results of a rat study. Physiol Meas. 2015 Oct;36(10):N115-26. doi: 10.1088/0967-3334/36/10/N115. Epub 2015 Sep 3. PMID 26334594
- [Background] Le Roux P, Menon DK, Citerio G, Vespa P, Bader MK, Brophy GM, Diringer MN, Stocchetti N, Videtta W, Armonda R, Badjatia N, Boesel J, Chesnut R, Chou S, Claassen J, Czosnyka M, De Georgia M, Figaji A, Fugate J, Helbok R, Horowitz D, Hutchinson P, Kumar M, McNett M, Miller C, Naidech A, Oddo M, Olson D, O'Phelan K, Provencio JJ, Puppo C, Riker R, Robertson C, Schmidt M, Taccone F; Neurocritical Care Society; European Society of Intensive Care Medicine. Consensus summary statement of the International Multidisciplinary Consensus Conference on Multimodality Monitoring in Neurocritical Care : a statement for healthcare professionals from the Neurocritical Care Society and the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Sep;40(9):1189-209. doi: 10.1007/s00134-014-3369-6. Epub 2014 Aug 20. PMID 25138226
- [Background] Harary M, Dolmans RGF, Gormley WB. Intracranial Pressure Monitoring-Review and Avenues for Development. Sensors (Basel). 2018 Feb 5;18(2):465. doi: 10.3390/s18020465. PMID 29401746
- [Background] Strandgaard S, Paulson OB. Cerebral autoregulation. Stroke. 1984 May-Jun;15(3):413-6. doi: 10.1161/01.str.15.3.413. No abstract available. PMID 6374982
- [Background] PEREZ-BORJA C, MEYER JS. A CRITICAL EVALUATION OF RHEOENCEPHALOGRAPHY IN CONTROL SUBJECTS AND IN PROVEN CASES OF CEREBROVASCULAR DISEASE. J Neurol Neurosurg Psychiatry. 1964 Feb;27(1):66-72. doi: 10.1136/jnnp.27.1.66. No abstract available. PMID 14123928
- [Background] Bodo M, Pearce FJ, Armonda RA. Cerebrovascular reactivity: rat studies in rheoencephalography. Physiol Meas. 2004 Dec;25(6):1371-84. doi: 10.1088/0967-3334/25/6/003. PMID 15712716
- [Background] Bodo M, Pearce FJ, Montgomery LD, Rosenthal M, Kubinyi G, Thuroczy G, Braisted J, Forcino D, Morrissette C, Nagy I. Measurement of brain electrical impedance: animal studies in rheoencephalography. Aviat Space Environ Med. 2003 May;74(5):506-11. PMID 12751577
- [Background] Bodo M, Pearce FJ, Baranyi L, Armonda RA. Changes in the intracranial rheoencephalogram at lower limit of cerebral blood flow autoregulation. Physiol Meas. 2005 Apr;26(2):S1-17. doi: 10.1088/0967-3334/26/2/001. Epub 2005 Mar 29. PMID 15798222
- [Background] Bodo M, Szebeni J, Baranyi L, Savay S, Pearce FJ, Alving CR, Bunger R. Cerebrovascular involvement in liposome-induced cardiopulmonary distress in pigs. J Liposome Res. 2005;15(1-2):3-14. doi: 10.1081/lpr-64523. PMID 16194924
- [Background] Armonda RA, Bell RS, Vo AH, Ling G, DeGraba TJ, Crandall B, Ecklund J, Campbell WW. Wartime traumatic cerebral vasospasm: recent review of combat casualties. Neurosurgery. 2006 Dec;59(6):1215-25; discussion 1225. doi: 10.1227/01.NEU.0000249190.46033.94. PMID 17277684
- [Background] Le Roux P, Menon DK, Citerio G, Vespa P, Bader MK, Brophy GM, Diringer MN, Stocchetti N, Videtta W, Armonda R, Badjatia N, Boesel J, Chesnut R, Chou S, Claassen J, Czosnyka M, De Georgia M, Figaji A, Fugate J, Helbok R, Horowitz D, Hutchinson P, Kumar M, McNett M, Miller C, Naidech A, Oddo M, Olson D, O'Phelan K, Provencio JJ, Puppo C, Riker R, Robertson C, Schmidt M, Taccone F. Consensus summary statement of the International Multidisciplinary Consensus Conference on Multimodality Monitoring in Neurocritical Care: a statement for healthcare professionals from the Neurocritical Care Society and the European Society of Intensive Care Medicine. Neurocrit Care. 2014 Dec;21 Suppl 2(Suppl 2):S1-26. doi: 10.1007/s12028-014-0041-5. PMID 25208678
- See also: ICM+ — http://www.neurosurg.cam.ac.uk/pages/ICM/about.php
- See also: Monitoring cerebrovascular pressure reactivity with rheoencephalography — https://doi.org/10.1088/1742-6596/224/1/012089
- See also: In vivo cerebral blood flow autoregulation studies using rheoencephalography — https://iopscience.iop.org/article/10.1088/1742-6596/224/1/012088